CLINICAL TRIAL: NCT04131764
Title: Utility of Quantification of Afferent Pupillary Defect in Predicting Optic Nerve Disease in Retrobulbar Neuritis, Multiple Sclerosis and Neuromyelitis Optica Spectrum Disease - a Retrospective and Prospective Analysis
Brief Title: Diagnosis of ON With or Without MS or NMOSD
Status: Terminated | Type: Observational
Why Stopped: IRB closed
Sponsor: Jagannadha R Avasarala (Other)
Responsible Party: Sponsor-Investigator, Jagannadha R Avasarala, Professor of Neurology, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 53342
Record Dates: First submitted 2019-10-17; First posted 2019-10-18 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorder Attack; Neuromyelitis Optica Spectrum Disorder Relapse; Neuromyelitis Optica Spectrum Disorder Progression; Optic Neuritis
Keywords: multiple sclerosis; MS; Neuromyelitis optica spectrum disorder; NMOSD; optic neuritis; pupillary response; RAPD; rapid afferent pupillary defect
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis; Neuromyelitis Optica | interventions — Reflex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Optic neuritis diagnosis only: Patients who have a diagnosis of optic neuritis, without a diagnosis of MS or NMOSD.
  Interventions: Diagnostic Test: Reflex (Brightlamp Inc., Purdue University)
- ON and multiple sclerosis: Patients who have a diagnosis of optic neuritis AND multiple sclerosis.
  Interventions: Diagnostic Test: Reflex (Brightlamp Inc., Purdue University)
- ON and NMOSD: Patients who have a diagnosis of optic neuritis and neuromyelitis optica spectrum disorder.
  Interventions: Diagnostic Test: Reflex (Brightlamp Inc., Purdue University)

INTERVENTIONS:
Diagnostic Test: Reflex (Brightlamp Inc., Purdue University) — The Reflex pupillometer is a mobile based application that provides a quantitative way to monitor pupillary activity and responsiveness. It uses the mobile phone as a source of light and records pupillary response, as well as analyzes and compiles the data. It produces quantitative measures such as latency, minimum and maximum pupil diameter, maximum and average constriction velocity, dilation velocity, and 75% recovery time.

SUMMARY:
This is both a prospective and retrospective study of patients with a known diagnosis of optic neuritis (ON) only, multiple sclerosis (MS) with ON, or neuromyelitis spectrum disorder (NMOSD) with ON. There will be no requirement for blinding (patient or assessor) and data collected with the Reflex app will be compared against other data that track optic nerve functional status, such as optical coherence tomography (OCT), visual fields (VF), low-contrast sensitivity, MRI orbits/brain and visual evoked potentials (VEP). Patients who have any diagnosis of ON, with or without a diagnosis of MS or NMOSD and who have had testing using other modalities such as VEPs, VF, low-contrast sensitivity studies, OCT, and MRI of brain or orbits will be included as retrospective subjects in the study. In this cohort, RAPD assessments will be completed and compared to against the data that has accrued as noted.

DETAILED DESCRIPTION:
The purpose of this research is to gather information on whether using quantitative- or numerical measurements of pupil changes as an alternative to qualitative- or observation based- testing can be done to assess optic nerve dysfunction in ON, MS with ON, and NMOSD with ON. One way this is done is through evaluating relative afferent pupillary defect (RAPD), which is a clinical sign that is used to detect an injury or defect in the pupil's pathway and this often involves the retina of the eye, which focuses light, and the optic nerve, which sends visual information to the brain. When shining a light into each eye, the eye with RAPD shows a slowed response to light, and when the light moves to the normal eye, the pupil of RAPD eye will dilate. Observational evaluations of RAPD are very common in clinical neurology to detect these optic nerve diseases. As technology has advanced, to lessen the observation errors, numerical measurement of RAPD is now possible through a web based app called Reflex (Brightlamp Inc., Purdue University), which is a FDAapproved class I regulated medical device. In this study, the investigator will compare the results of a participant's app recording to other data that has been collected which also tracks optic nerve function status.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ages 18-90 years
2. Signed informed consent
3. Have been diagnosed with optic neuritis (ON) only, MS and ON, or NMOSD and ON
4. Have had at least one previous test to track optical nerve function

Exclusion Criteria:

1. Are pregnant or nursing
2. Are children (age <18 years)
3. Do not have a diagnosis of optic neuritis (ON)
4. Have a diagnosis of MS or NMOSD without a diagnosis of ON as well

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients include those seen at the University of Kentucky during routine clinical neurology visits between the ages of 18 and 90 years who have been diagnosed with optic neuritis, optic neuritis and multiple sclerosis, or optic neuritis and neuromyelitis optica spectrum disorder and have had at least one previous test that tracks optic nerve function.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of device for diagnosis of ON | 10 seconds
  Feasibility of using quantified pupillary responses as a surrogate marker for assessment of optic nerve dysfunction in ON, MS, and NMOSD.
Comparative data assessment | Time of app scan (10s) plus time to compare data (1-2 hours)
  Comparing Reflex with other routine clinical methods of evaluating optic nerve dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Jagannadha Avasarala, MD PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Reflex User Guide — https://static1.squarespace.com/static/5c269669297114a6e7a6cf31/t/5c658ae0652dea8b1f6b4b72/1550158561852/Reflex+User+Guide.pdf